CLINICAL TRIAL: NCT05943600
Title: An Assessment of Treatment Adherence of Osteoporosis Patients From a Biopsychosocial Perspective to Plan a Multidisciplinary Intervention Overcame Psychosocial Barriers
Brief Title: An Assessment of Treatment Adherence of Osteoporosis Patients From a Biopsychosocial Perspective
Status: Not yet recruiting | Type: Observational
Sponsor: Istanbul University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Esin Temeloglu Sen, Research Assistant Dr. (PhD), Istanbul University
Other Study IDs: OPKO-1
Record Dates: First submitted 2023-06-13; First posted 2023-07-13 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: Osteoporosis; Osteoporotic Fractures; Psychosocial Functioning; Medication Adherence
Keywords: osteoporosis; fragile fracture risk; medication adherence; psychological symptom level; biopsychosocial model
MeSH Terms: conditions — Osteoporosis; Osteoporotic Fractures; Medication Adherence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Osteoporosis patients: Participants will fill out the self-report scales.

SUMMARY:
This observational study aims to learn about the psychosocial risk factors of osteoporosis (OP) patients. The main question it aims to answer is:

* Which biopsychosocial factors affect OP patients' fragility fracture risk regarding the health behaviour model? Participants will fulfil these forms below here;
* Sociodemographic and Clinical Information Form,
* Fragility Fracture Information Form
* Medication Adherence Report Scale
* Brief Illness Perception Scale
* The Beliefs About the Medicines Scale-Specific
* The Short Assessment of Patient Satisfaction
* Perceived Stress Scale
* Multidimensional Perceived Social Support Scale
* Brief Symptom Inventory - Depression and Anxiety
* Health Behavior Assessment Scale

DETAILED DESCRIPTION:
Osteoporosis (OP) is a disease characterized by decreased bone density and deterioration of bone microarchitecture. Fracture risk, which is one of the most negative disease experiences faced by OP patients, can be seen in many parts of the body in the later stages of the disease. The necessity of interventions that prevent or delay fractures highlights severe orthopaedic surgeries, increasing health expenditures and psychosocial losses in the lives of individuals. The project will proceed through three objectives: researching the components that affect the fracture, developing an intervention and implementing it. According to the first aim, it has been seen in the current literature that the most effective method in preventing the risk of fracture is to increase the medication adherence (MA) of the patients. It is seen that the Self-Regulatory Model (SRM)-based studies, in which the components explaining the MA of OP patients are examined as a model, constitute one of the limited theory-based studies. However, the SRM, which stands out as an effective model in explaining MA with its components of "perception of illness" and "beliefs about the medicine", is thought to base the medication use experience only on individual validities. Hence, the concept of MA is also provided by the patient-doctor relationship. Therefore, the effect of patient satisfaction on MA will be discussed in the components of SRM. There are also psychosocial factors that are thought to affect the possible fracture apart from all these diseases and treatment-related components. There are findings that the fear of falling, anxiety and social withdrawal caused by OP increase the risk of a possible fracture. Accordingly, patients' psychological challenges may affect protective behaviours such as exercise and a calcium-rich diet, and smoking. Therefore, it is predicted that the psychological symptom levels of the patients will affect the fracture through health behaviours. Besides, OP can bring along stress just like other chronic diseases, and perhaps even more social support needs can be seen in these patient groups with other chronic diseases. Hence, the moderator effect of social support between the psychological symptom level of OP patients and their stress' constitutes another sub-research question of this study. It is aimed to develop a comprehensive multidisciplinary and evidence-based intervention that prevents possible fracture experiences in OP patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary or secondary osteoporosis or osteopenia with a previous fragility fracture
* Taking osteoporosis medicines for at least 6 months
* Volunteer to attend to study

Exclusion Criteria:

* Having been diagnosed with osteoporosis for less than six months
* Not willing to fulfil the requirements of the study
* Having a neurological (such as dementia) or psychological (such as psychosis) condition that prevents completing the scales and establishing a relationship with the tester.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Osteoporosis patients take for at 6 months.
Sampling Method: Non-Probability Sample
Enrollment: 585 (Estimated)
Dates: Start 2023-07-15 (Estimated); Primary Completion 2024-03-15 (Estimated); Study Completion 2026-04-15 (Estimated)

PRIMARY OUTCOMES:
Medication Adherence Report Scale | through study completion; approximately 9 months
  This scale will be used to assess the medication adherence level of patients. The scale is scored between 5 to 25 points with lower scores indicating higher adherence level.
Fragility Fracture Information Form | through study completion; approximately 9 months
  The form will be used to assess the fragility fracture experience of participants. There are no cut-off values since this form will give the investigators descriptive information.
Health Behavior Assessment Form | through study completion; approximately 9 months
  The form will be used to assess the smoking, diet or alcohol consumption of participants. There are no cut-off values since this form will give the investigators descriptive information.

SECONDARY OUTCOMES:
Brief Illness Perception Scale | through study completion; approximately 9 months
  The scale will be used to assess participants' illness perception and cognition. To score the Brief Illness Perception Scale questionnaire, each item is rated on a 0-10 scale, with higher scores indicating a more threatening perception of the illness. The total score is calculated by summing the scores of all seven items, with a possible range of 0-70. Higher scores indicate worse illness perception.
The Beliefs About the Medicines Scale-Specific | through study completion; approximately 9 months
  The scale will be used to assess the appraisal of the medicines. The Beliefs About the Medicines Scale-Specific consists of two five-item scales assessing participants' beliefs about the necessity of prescribed medication for controlling their disease and their concerns about potential adverse consequences of taking it. Respondents indicate their degree of agreement with each statement on a five-point Likert scale, ranging from 1=strongly disagree to 5=strongly agree. Scores obtained for individual items within both scales are summed. A mean score for each scale is computed by dividing total scores for that scale by the number of items in the scale, resulting in a mean score range of 1-5 for each scale. Higher scores indicate stronger beliefs in the concepts represented by the scale.
The Short Assessment of Patient Satisfaction | through study completion; approximately 9 months
  The scale will be used to assess patient satisfaction comprised of a short seven-item scale that has 5-point responses, scored as 0 to 4. The scale assesses the core domains of patient satisfaction which includes treatment satisfaction, explanation of treatment results, clinician care, participation in medical decision-making, respect by the clinician, time with the clinician, and satisfaction with clinic care. The score ranges from 0 (extremely dissatisfied) to 28 (extremely satisfied), as a continuous score. Additionally, categorical scores are defined as 0-10 very dissatisfied, 11-18 dissatisfied, 19-26 satisfied, and 27-28 very satisfied.
Perceived Stress Scale | through study completion; approximately 9 months
  The scale will be used to assess the stress perception of participants. The scores on the Perceived Stress Scale can range from 0 to 40 with higher scores indicating higher perceived stress. Scores ranging from 0-13 would be considered low stress; scores ranging from 14-26 would be considered moderate stress, and scores ranging from 27-40 would be considered high perceived stress.
Multidimensional Perceived Social Support Scale | through study completion; approximately 9 months
  The scale will be used to assess the social support level of participants. The scale is a short instrument designed to measure an individual's perception of support from 3 sources: family, friends and a significant other. To calculate the total score, all 12 items are summed. This total score can also be calculated as a mean score (dividing by 12). A mean scale score ranging from 1 to 2.9 could be considered low support; a score of 3 to 5 could be considered moderate support; a score from 5.1 to 7 could be considered high support.
Brief Symptom Inventory- Depression and Anxiety | through study completion; approximately 9 months
  The scale is a 13-item self-report scale designed to evaluate the depression and anxiety symptoms levels of participants. This scale uses a 5-point Likert scale, ranging from 0 ("not at all") to 4 ("extremely"). Brief Symptom Inventory- Depression and Anxiety scores can range from 0 to 52 points with higher scores indicating higher suffering from depression and anxiety symptoms.

OTHER OUTCOMES:
Sociodemographic and Clinical Information Form, | through study completion; approximately 9 months
  The form will be used to get an illness history and demographical information. There are no cut-off values since this form will give the investigators descriptive information.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University, Istanbul Faculty of Medicine, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
We will not share any individual participant data with other researchers.

REFERENCES:
- [Background] Clyne W, Mshelia C, McLachlan S, Jones P, de Geest S, Ruppar T, Siebens K, Dobbels F, Kardas P. A multinational cross-sectional survey of the management of patient medication adherence by European healthcare professionals. BMJ Open. 2016 Feb 1;6(2):e009610. doi: 10.1136/bmjopen-2015-009610. PMID 26832430
- [Background] Chandran M, Tan MZ, Cheen M, Tan SB, Leong M, Lau TC. Secondary prevention of osteoporotic fractures--an "OPTIMAL" model of care from Singapore. Osteoporos Int. 2013 Nov;24(11):2809-17. doi: 10.1007/s00198-013-2368-8. Epub 2013 Apr 25. PMID 23615816
- See also: Medication adherence project final report — http://abcproject.eu/index.php?page=publications